CLINICAL TRIAL: NCT02007330
Title: The Effect of Systemic Lidocaine Infusion to Postoperative Pain and Quality of Recovery After Laparoscopic Hernia Repair in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2013-0692
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Inguinal Hernia
Keywords: systemic lidocaine; postoperative pain; recovery, pediatric; inguinal hernia; laparoscopy
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group L (Experimental): Intravenous lidocaine infusion group
  Interventions: Drug: Systemic intravenous lidocaine infusion
- Group C (Placebo Comparator): Intravenous normal saline infusion - control group
  Interventions: Drug: Normal saline infusion

INTERVENTIONS:
Drug: Systemic intravenous lidocaine infusion — In group L, intravenous lidocaine infusion (0.1mg/kg) for 1minutes after induction of anesthesia. After 1 minutes, lidocaine infusion continued at rate of 1.5mg/kg/hr during operation, and discontinued before move the patients to PACU.
  Arms: Group L
Drug: Normal saline infusion — In group C, the patients receive same volume of normal saline
  Arms: Group C

SUMMARY:
Systemic lidocaine administration may improve postoperative pain and recovery after laparoscopic inguinal hernia repair in pediatric patients

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 and 6 year-old
* ASA class 1 and 2
* Pediatric Inguinal hernia patients who are scheduled for elective laparoscopic inguinal hernia repair

Exclusion Criteria:

* Allergy to local anesthetics or contraindication to use of lidocaine
* Current active upper respiratory infection or history of upper respiratory infection within 2 weeks
* Severe cardiovascular disease
* Renal failure
* Liver failure
* Neurologic and psychologic disease
* Chronic treatment with analgesics
* Previous history of laparoscopic operation
* Parents' refusal

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Assessing postoperative pain | 24 hours after operation
  Assessing FLACC(Face-Legs-Activity-Crying-Consolability) score at 4, 8, 12 and 24hours after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea